CLINICAL TRIAL: NCT02097836
Title: Segmental Training for Trunk Control a Pilot Study for Children With Moderate to Severe Motor Impairment.
Brief Title: Targeted Training for Trunk Control_case Series Cerebral Palsy
Acronym: CP_TT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP_TT_2008
Record Dates: First submitted 2014-03-24; First posted 2014-03-27 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Cerebral Palsy; Traumatic Brain Injury
Keywords: postural control; Targeted Training; cerebral palsy; trunk segments
MeSH Terms: conditions — Cerebral Palsy; Brain Injuries, Traumatic

STUDY DESIGN:
Masking Description: Gross Motor Function Measure Outcome was masked for temporal order and video scored by reviewers who were not involved in data collections or intervention.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single subject case series (Experimental): Targeted training, 5-6 days a week for 6 months, minimum of 20 minutes per day
  Interventions: Device: Targeted Training

INTERVENTIONS:
Device: Targeted Training — Custom training devices were imported from The Movement Centre for research purposes. The typical course of treatment involves loaning the customized equipment to each family for use in their home or in their child's educational setting. Training occurs once daily usually for 30-45 minutes. This is done 5 or 6 days per week. Training programs typically involve playing with balls or balloons or video games that motivate the child to hold the head erect and to wave the arms and hands and move the upper body.

SUMMARY:
If a child with cerebral palsy does not develop independent sitting balance by 4 years of age, their prognosis for walking is very poor. Surprisingly little is known about how to facilitate head control or upright sitting balance and functional mobility in the child who is not developing these skills. This is one of the first studies that will examine intermediate stages in the development of the postural control system in children with neurologic deficits. Clinical researchers at The Movement Centre in Oswestry, England have developed a method called Targeted Training in which trunk control is trained in children segment by segment using a specific training device. This study aims to examine kinematic and electromyographic changes in a case series of children who undergo a 6-month Targeted Training intervention.

ELIGIBILITY:
Inclusion Criteria:

* neurologic diagnosis that results in a deficit in trunk control (i.e. cerebral palsy, traumatic brain injury)
* age 4-17 years
* Gross Motor Function Classification System (GMFCS) level III, IV or V for children with cerebral palsy

Exclusion Criteria:

* spinal fixation
* fixed scoliosis
* uncontrolled seizures

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2007-09; Primary Completion 2009-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Change in Gross Motor Function Measure | 6 months and followup post training 12 months
Probe data, balance | baseline, intervention, 2 months post intervention
  timed balance task

SECONDARY OUTCOMES:
Change in head stability | 6 months, 1,3, and 12 months post intervention
  Change in alignment and stability of head postural sway during quiet sitting
Change in muscle activation strategy during quiet sitting with different levels of external support. | 6 months, 1 and 3 months post intervention
Change in Pediatric Evaluation of Disability Inventory (PEDI) | 6 months and 1,3, 12 months post intervention
Qualitative Parent, Teacher report | during intervention and post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sandra L Saavedra, PhD, Principal Investigator — University of Oregon